CLINICAL TRIAL: NCT00144859
Title: A 28-day, Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Anti-inflammatory Effect and Steady-state Pharmacokinetics of SB-681323 7.5 mg Per Day in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Safety And Anti-Inflammatory Effect Of SB681323 In Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKC101614
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: P38 map kinase; CRP; COPD; safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dilmapimod

INTERVENTIONS:
Drug: SB681323

SUMMARY:
This is a 28-day, placebo controlled clinical study assessing the safety, tolerability anti-inflammatory effect and pharmacokinetics of SB681323 in patients with COPD (Chronic Obstructive Pulmonary Disease).

ELIGIBILITY:
Inclusion criteria:

* Non-childbearing potential.
* Clinical diagnosis of COPD.
* Cigarette smoking history of greater than or equal to 10 pack years.
* Post-bronchodilator FEV1 to FVC ratio (FEV1:FVC) < 0.7
* Post-bronchodilator FEV1 50% - 80% of predicted normal.
* Receiving inhaled corticosteroids for a minimum of 6 weeks prior to Screening.
* Serum CRP concentration greater than 3mg/L.

Exclusion criteria:

* Current diagnosis of asthma.
* Active tuberculosis, sarcoidosis or bronchiectasis.
* History of any type of malignancy, rheumatoid arthritis or other conditions associated with chronic inflammation.
* Clinically significant renal or hepatic disease.
* History of increased liver function tests, or patients receiving hormone replacement therapy, statins or systemic or topical corticosteroids.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 2005-07

PRIMARY OUTCOMES:
Safety and tolerability as assessed by incidence of elevated liver function tests. Serum concentration c-reactive protein (CRP)

SECONDARY OUTCOMES:
Inflammatory markers in blood and sputum Spirometric lung function tests Dyspnoea measured by the TDI Safety assessments Population Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Denmark (2):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, København NV
- GSK Investigational Site, Helsinki, Finland
- Germany (4):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- Netherlands (4):
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- United Kingdom (6):
  - GSK Investigational Site, Liverpool, Lancashire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London